CLINICAL TRIAL: NCT02992795
Title: A Study to Assess the Effectiveness of the BrainPulse as an Aid to the Diagnosis of Concussion
Brief Title: Unblinded Data Collection Study of Concussion Using BrainPulse
Status: Completed | Type: Observational
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JMC-1602
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Concussion, Intermediate
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Cohort Ia: Athletes in this cohort serve as control subjects participating in Division 1 Athletics at the University of Wyoming. They will be enrolled once they meet eligibility. Upon enrollment, all athletes will have an initial BrainPulse recording. Once a subject from this cohort sustains an injury, they crossover to Cohort II. Also, a matched control for every concussed subject will be selected from Cohort Ia.
  Interventions: Device: BrainPulse
- Cohort Ib: Athletes in this cohort are subjects currently subscribed to the Head Health Network. They will have a BrainPulse recording completed every week through the entire season. Similarly, if subjects in this cohort sustain an injury, they will crossover to Cohort II.
  Interventions: Device: BrainPulse
- Cohort IIa: Athletes from Cohort I will be assigned to cohort IIa once they sustain an injury other than concussion. They will have been pulled out of the game by the athletic trainer and removed from play until at least the end of the game. Once the subjects have been assigned to Cohort IIa, they will have a BrainPulse recording and a symptom evaluation within 3 days of their injury. After two weeks of recovery, subjects in this cohort will return to Cohort 1 and resume their participation in the study in their respective sub-cohort.
  Interventions: Device: BrainPulse
- Cohort IIb: Athletes in this cohort are injured subjects who sustain a non-penetrating head injury and are confirmed to have had a concussion according to the protocol reference standard and by their physician. All subjects enrolled in this cohort are required to have a BrainPulse recording within 3 days of their injury. Each BrainPulse recording will be accompanied by a symptoms evaluation and medical data collection documented in the case report forms. Subjects will complete 3 weeks of follow-up visits post injury.
  Interventions: Device: BrainPulse

INTERVENTIONS:
Device: BrainPulse — JanMedical's BrainPulse measures the brain motion caused by pulsatile blood flow from the cardiac cycle referred to as the BrainPulse signal. The BrainPulse measures skull acceleration in response to tge brain motion using an array of sensors placed on the head.

SUMMARY:
This is a prospective, non-blinded, matched control study of young athletes (ages 10-28 years old) in collegiate sports. The cohorts are defined in accordance to the athlete's exposure of injury. All subjects will complete a minimum of one recording based on their assigned cohort. Concussed athletes will complete an additional 3 weeks of follow-up recordings post injury. The symptomatic evaluation, physical examination, neurological baseline testing, and BrainPulse recordings will be entered in a database to determine clinical outcome and assess device utilization.

DETAILED DESCRIPTION:
Cohort I is defined as all enrolled athletes at the University of Wyoming and is divided into two sub-cohorts: Cohort Ia include all athletes participating in Division 1 Athletics; Cohort Ib are athletes subscribed to the Head Health Network. Cohort II is defined as all injured athletes participating in the teams and includes two sub-cohorts: Cohort IIa is defined as non- concussed injured athletes; Cohort IIb concussed athletes per reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female young athletes between ages 18-28 yrs
2. Enrolled at the University of Wyoming and currently participating in Division 1 Athletics
3. Completed the following baseline testing: SWAY balance, King-Devick, C3-Logix
4. Willing and able to participate in all study evaluations and allow access to medical testing and records
5. Signed informed consent, or have a legally authorized representative willing to provide informed consent on behalf of the subject if the subject is a minor

Exclusion Criteria:

1. Prior concussion diagnosed by a physician in the last 2 weeks assessed via interview with athlete (not including a recent concussion within the last 3 days)
2. Any serious medical, social or psychological condition that in the opinion of the investigator would impair ability to provide informed consent or otherwise disqualify a patient from participation

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletes participating in Division 1 Athletics at the University of Wyoming
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Comparison of BrainPulse recordings of concussed subjects with BrainPulse recordings from their matched Controls | Through study completion, expected to be 8 months
  Collect BrainPulse data from at least 15 concussed athletes and matched controls to develop and improve algorithms that can aid in the diagnosis of concussion.
  The specific signal patterns observed from confirmed concussed subjects' BrainPulse recordings will be evaluated against the BrainPulse recordings from the matched control subjects.

SECONDARY OUTCOMES:
Correlate helmet sensor's force of impact measurements with BrainPulse data | Through study completion, expected to be 8 months
  Compare the magnitude of force measured by helmet sensors from subconcussive hits with consecutive BrainPulse recordings. As such, BrainPulse data on these athletes will be compared with helmet sensor data, baseline cognitive testing, and the initial BrainPulse recording.
Compare BrainPulse Data between Injured Athletes, Non-Injured athletes, and Concussed Athletes | Through study completion, expected 8 months
  Compare BrainPulse signals in subjects sustaining a non-concussive injury to subjects that have a confirmed diagnosis of concussion. Also compare BrainPulse signals from injured subjects in Cohort IIa with non-injured subjects in Cohort Ia.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No
All study outcome measures will be made available within 6 months of study completion